CLINICAL TRIAL: NCT05847452
Title: Beyond the Eosinophil: Understanding the Impact of Eosinophil Depletion on T2 Inflammation. (BEUTI)
Acronym: BEUTI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 310865
Record Dates: First submitted 2023-04-03; First posted 2023-05-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: Asthma; Benralizumab
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/ plasma/ cells (blood) Airway samples: Endobronchial biopsy (small lung tissue pieces), bronchial brushings (contains bronchial epithelial cells) bronchoalveolar lavage (fluid and cells collected from the lungs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All eligible participants will be consented and enrolled into the study and given the IMP as follows:
  Benzraliziumab 30mcg once a month for 3 months
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — 30mcg ever month for 3 months

SUMMARY:
Benralizumab is a relatively new treatment that is approved by NICE (National Institute for Health and Care Excellence, https://www.nice.org.uk/) for patients with severe asthma who have ongoing eosinophilic inflammation that remains poorly controlled despite high dose inhaled glucocorticosteroid medication.

Eosinophils are a type of white blood cell that are linked to allergy and inflammation and are raised in people with severe asthma. Severe asthma is associated with a type-2 (T2) inflammation phenotype characterised by increased T2 cytokines (IL-13, IL-4, IL-5). Increased levels of eosinophils can cause inflammation in the lungs, increasing the risk of asthma attacks. The standard treatment for asthma involves taking inhaled glucocorticosteroid medication which primarily work by suppressing eosinophilic inflammation in the lungs.

Benralizumab is a monoclonal antibody that targets a receptor on the surface of eosinophils called interleukin-5 receptor-α (IL-5Rα) leading to the rapid death of these cells and consequently a reduction in airways inflammation.

In clinical trials, benralizumab has been shown to reduce both symptoms and the number of asthma attacks suffered by those with severe eosinophilic asthma. However, it remains unclear whether this clinical efficacy relates purely to the removal of the eosinophil, or additionally to the impact of this on other parts of the immune system.

The BEUTI study will examine the structure and function of airway cells in patients with severe eosinophilic asthma. Particularly how the immune function of these cells changes with treatment and whether benralizumab leads to a reduction in T2 mediators and/or activation in airway cells.

The aim is to take samples of cells from the airways during a bronchoscopy (a camera test looking into the lungs) before starting benralizumab and after 12 weeks of treatment. These investigations will allow us to better understand how benralizumab affects the cells within the airways and the pathways involved.

DETAILED DESCRIPTION:
Benralizumab is a relatively new treatment that is approved by NICE for patients with severe asthma and ongoing eosinophilic inflammation that remains poorly controlled despite high dose inhaled corticosteroid medication. Benralizumab targets a receptor on the surface of eosinophils called IL-5R leading to the rapid death of these cells and consequently a reduction in airways inflammation. In clinical trials, benralizumab has been shown to reduce both symptoms and the number of asthma attacks suffered by those with severe eosinophilic asthma. However, it remains unclear whether this clinical efficacy relates purely to the removal of the eosinophil, or additionally to the impact of this on other parts of the immune system including activation of type-2 (T2) inflammation pathways.

The clinical effectiveness of benralizumab is evident across phase 3 and real world studies which has reaffirmed the central role that the eosinophil plays in disease and exacerbation pathogenesis in patients with severe asthma. However, whilst it is generally believed that this fundamentally reflects the removal of eosinophils and their toxic granules and mediators from the airway, the full impact of benralizumab on T2 immunity may be much broader.

Firstly, benralizumab-treated patients stop exacerbating when they encounter respiratory viruses such as rhinovirus, suggesting that the deficient anti-viral immune responses present in many uncontrolled T2-high asthmatics are restored upon benralizumab. Secondly, our centres' finding that patients continue to remain well-controlled despite significantly reducing their inhaled corticosteroid (ICS) use following initiation of benralizumab suggests that the other elements of T2 inflammation (including IL-13 driven pathways) are either unimportant or suppressed (d'Ancona et al., Allergy 2021, vol; 76(7):2238-2241). Thirdly our observation that benralizumab is very effective in patients with high fractional exhaled nitric oxide (FeNO) levels (indicating increased IL-13-driven activation) and that treatment significantly reduces FeNO levels suggests that benralizumab directly or indirectly suppresses IL-13 pathways (Hearn et al., J Allergy Clin Immunol Pract, 2021, Vol;9(5):2093-2096). Taken together, there is an increasing body of data supporting the notion that benralizumab has far-reaching anti-T2 effects that underpin its excellent efficacy in clinical practice. Through the use of novel techniques including spatial transcriptomics of bronchial biopsies this proposal aims to define and describe these effects.

Study Hypothesis:

The depletion of eosinophils by benralizumab leads to additional inhibitory effects on T2 inflammation which collectively underpins the improvements in multiple clinical domains and reduction in T2 biomarkers observed in real world cohort studies.

The important research questions we will aim to answer:

i) What is the effect of benralizumab on T2 signalling. Can benralizumab modulate T2-signalling and/or gene expression in addition to triggering eosinophil and basophil depletion? ii) What additional cell types (e.g. ILC2, alveolar macrophages, mast cells, bronchial epithelial cells, airway smooth muscle) are regulated by benralizumab? iii) Does the marked reduction in exacerbations observed with benralizumab partly reflect restoration of the deficient anti-viral immune responses seen in patients with severe asthma?

The investigators plan to take samples of cells from the airways during a bronchoscopy (a camera test looking into the lungs) before starting benralizumab and after 12 weeks of treatment. These investigations will allow us to better understand how benralizumab affects the cells within the airways.

BEUTI study primary objective is to investigate the impact of benralizumab treatment on lung inflammation and airway structure in patients with severe eosinophilic asthma. Its secondary objective is to understand if benralizumab treatment affects response to infection with respiratory viruses such as the common cold virus (rhinovirus) and SARS CoV2.

Benralizumab will be commenced according to UK NICE severe asthma guidance with 30mg sub cutaneous dosing every 4 weeks for first 3 doses, followed by every 8 weeks.

The BEUTI study will have a total of 8 visits with 2 bronchoscopies (to collect airway cells and blood cells) at visit 2 and visit 8.

Throughout the study, information regarding their asthma symptoms, adverse events and lung function will be collected.

Asthma control score and quality of life questionaire (ACQ-6/mAQLQ). Breathing tests will be performed (spirometry, fractional exhaled nitric oxide (FeNO)).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Patients aged 18 and over with a diagnosis of severe eosinophilic asthma for at least the last 6 months
3. Eligible for benralizumab based on NICE criteria
4. Poorly-controlled (ACQ-6 >1.5)
5. FeNO ≥50ppb at screening despite high dose inhaled corticosteroids (at least 1000mcg BDP equivalent) +/- maintenance prednisolone
6. Adult-onset (18+) asthma in a minimum of 50% of the study subjects

Exclusion Criteria:

1. Other severe eosinophilic lung disease including EGPA, chronic eosinophilic pneumonia and ABPA
2. Maintenance daily oral corticosteroids (prednisolone)
3. Severe bronchiectasis on CT causing daily sputum production
4. Inability to give written informed consent
5. Current smoking or >20 pack year smoking history
6. Resting oxygen saturations <94% on air
7. Any severe cardiac or other non-asthma related co-morbidity that would make bronchoscopy and/or sedation high risk
8. Symptoms suggestive of a respiratory viral / bacterial infection within the last 3 weeks
9. Acute exacerbations of asthma requiring high dose prednisolone within the last 3 weeks
10. A change in dose of maintenance inhaled and/or oral corticosteroid dose within the last 3 weeks
11. Positive strongyloides serology following screening
12. Pregnancy or lactation
13. Hypersensitivity to benralizumab or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with poorly-controlled severe eosinophilic asthma who meet NICE criteria to commence biologic therapy with benralizumab.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The change in the number of inflammatory cells in patients with severe eosinophilic asthma at baseline and after 12 weeks of benralizumab treatment. | 12 weeks
  To investigate the changes in the number of inflammatory cells in patients with severe eosinophilic asthma at baseline and after 12 weeks of benralizumab treatment.
The change in the activation status of Type-2 related cells in patients with severe eosinophilic asthma at baseline and after 12 weeks of benralizumab treatment. | 12 weeks
  Activation status will be measured by the relative expression of Type 2 inflammatory cells and gene expression

SECONDARY OUTCOMES:
To investigate changes in epithelial barrier integrity using transepithelial resistance before and after completing treatment with 12 weeks of benralizumab. | 12 weeks
  Transepithelial resistance measures changes in voltage across epithelial cells
To investigate changes in epithelial antiviral responses in untreated vs respiratory virus-infected cells including rhinovirus-16 in epithelial cells collected before and after completing 12 weeks of treatment. | 12 weeks
  Gene expression will be measured using RNA sequencing and reported as gene counts
To investigate changes in antiviral responses of alveolar macrophages to respiratory viruses including rhinovirus-16 in cells collected from the airways before and after completing 12 weeks of treatment. | 12 weeks
  To investigate changes in antiviral responses of alveolar macrophages to respiratory viruses including rhinovirus-16 in cells collected from the airways before and after completing 12 weeks of treatment using protein and nucleic acid analyses.
To investigate changes in epithelial responses to pro-inflammatory cytokines/chemokines in cells collected before and after treatment. | 12 weeks
  To investigate changes in epithelial responses to pro-inflammatory cytokines/chemokines in cells collected at baseline and after treatment.
To investigate changes in Type 2 inflammation in peripheral airways by collecting bronchoalveolar lavage fluid before and after treatment for nucleic acid and protein analyses. | 12 weeks
  Change in the cellular proportions of Type 2 inflammatory cells will be measured using RNA sequencing and reported as gene counts
To investigate changes in peripheral airway dysfunction before and after treatment by measuring impulse oscillometry. | 12 weeks
  Impulse oscillometry will be measured as resistance and impedance
To investigate the change in FeNO levels before and after treatment. | 12 weeks
  FeNO will be measured in parts per billion (ppb)
Change in routine full blood counts including eosinophil and basophil numbers. | Regular timepoints during 12 weeks
  Change in routine full blood counts including eosinophil and basophil numbers at baseline and following 12 weeks of treatment.
Asthma control measured by Asthma Control Questionnaire (ACQ)-6 | 12 weeks
  Asthma control questionnaire completed at baseline and following 12 weeks of treatment. Total score ranges from 0-6, with 0=no impairment due to asthma, 6 = maximum impairment due to asthma.
Quality of Life Score measured by the mini Asthma Quality of Life Questionnaire (mAQLQ) | 12 weeks
  Change in mAQLQ score at baseline and following 12 weeks of treatment. Score for each question ranges from 0-7, with 0 = totally limited, 7 = not limited at all. The score is calculated as an average for each domain, with a clinically minimum difference of 0.5.
Change in lung function parameters measured by spirometry (FEV1, FVC, FEV1/FVC) | 12 weeks
  Change in lung function parameters at baseline and after 12 weeks of treatment measured by spirometry (FEV1, FVC, FEV1/FVC)
Change in the number of airway immune cells and their activation status as well as spatial location in endobronchial biopsies as measured by immunohistochemistry and spatial transcriptomic methods. | 12 weeks
  Change in the number of airway immune cells and their activation status as well as spatial location in endobronchial biopsies as measured by immunohistochemistry and spatial transcriptomic methods.
Change in airway remodelling by assessing structural cells (such as fibroblasts and smooth muscle) using immunostaining and histological examination | 12 weeks
  Change in airway remodelling by assessing structural cells (such as fibroblasts and smooth muscle) using immunostaining and histological examination

CONTACTS AND LOCATIONS:
Overall Officials: Prof. David Jackson, PhD, Principal Investigator — Guy's and St. Thomas NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT05847452/Prot_000.pdf